CLINICAL TRIAL: NCT05684146
Title: Protect the Head to Head: A Safety and Efficacy Assessment of the Emboliner Embolic Protection Device
Brief Title: Protect the Head to Head Study
Acronym: ProtectH2H
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Emboline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP-0527
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-01

CONDITIONS: Embolism
Keywords: MACCE; TAVR; Embolism
MeSH Terms: conditions — Embolism | interventions — Embolic Protection Devices

STUDY DESIGN:
Intervention Model Description: G4: Model Description* Subjects will be randomized (1:1) to either the Emboliner (ARM 1) or Sentinel CPS (ARM 2). Device randomization will be stratified by (a) site and (b) TAVR device type (Edwards or Medtronic) to ensure that each study arm represents an equivalent patient population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Emboliner Embolic Protection Device (Experimental): Emboliner embolic protection device to be used during TAVR procedures for stroke prevention
  Interventions: Device: Emboliner Embolic Protection
- Sentinel Cerebral Protection System (Active Comparator): Sentinel Cerebral Protection System to be used during TAVR procedures for stroke prevention
  Interventions: Device: Sentinel Cerebral Protection

INTERVENTIONS:
Device: Emboliner Embolic Protection — Emboliner Embolic Protection Device will be used to capture and remove embolic material during transcatheter aortic valve replacement (TAVR) interventions
  Other Names: Embolic protection
  Arms: Emboliner Embolic Protection Device
Device: Sentinel Cerebral Protection — The Sentinel Cerebral Protection System will be used to capture and remove embolic material during transcatheter aortic valve replacement (TAVR) interventions
  Other Names: Embolic protection
  Arms: Sentinel Cerebral Protection System

SUMMARY:
Prospective, randomized, open label, multicenter, 2-arm, safety and efficacy study

DETAILED DESCRIPTION:
Prospective, randomized, open label, multicenter, 2-arm, safety and efficacy study to demonstrate safety and effectiveness based on non-inferiority of the study device (Emboliner EPD) compared to the control device (Sentinel CPS) in terms of a 30-day composite major adverse cardiac and cerebrovascular events (MACCE) rate - defined as all death, stroke and Stage 3 acute kidney injury - evaluated on a per-patient basis, post-TAVR procedures

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for treatment for symptomatic severe aortic stenosis using a FDA-approved TAVR valve according to current guidelines
2. Consented to the TAVR procedure
3. Subject and physician agree that subject will return for required post-procedure follow-up
4. Willing to participate in study and provide signed EC/IRB-approved informed consent
5. Eighteen (18) years or older at the time of consent

Exclusion Criteria:

1. Not undergoing a planned TAVR via transfemoral access
2. Severe allergy or hypersensitivity to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, nitinol, and/or contrast agents that cannot be pre-medicated
3. Uncorrected bleeding disorder
4. Hypercoagulation status that cannot be corrected by additional peri-procedural heparin
5. Myocardial infarction (MI) diagnosis <30 days prior to study procedure
6. History of substance abuse that may cause non-compliance with the protocol or confound the data interpretation
7. Cardiogenic shock, hemodynamic instability requiring inotropic support or mechanical heart assistance, or severe hypotension (systolic blood pressure <90 mmHg) at time of screening
8. History of a stroke < 180 days prior to study procedure
9. Active peptic ulcer or history of upper gastrointestinal (GI) bleeding < 90 days prior to study procedure
10. Congenital unicuspid aortic valve
11. Porcelain aorta, asymmetrical or sharp aortic calcifications, severe aortic tortuosity, shaggy aorta or mobile atheroma in the arch
12. Pre-existing prosthetic heart valve in any position, prosthetic ring, or severe (greater than 3+) mitral insufficiency
13. Current leukopenia, acute anemia, thrombocytopenia, history of chronic bleeding diathesis, or coagulopathy that requires treatment
14. Hypertrophic cardiomyopathy with or without obstruction
15. Left ventricular ejection fraction (LVEF) ≤20%
16. Echocardiographic evidence of intracardiac or aortic mass, thrombus, or vegetation
17. Active infection or endocarditis
18. Neurodegenerative or other progressive neurological disease or history of significant head trauma followed by persistent neurologic defaults
19. Carotid stent placement or endarterectomy performed <180 days prior to study procedure.
20. Severe renal insufficiency (creatinine >3.0 mg/dL or GFR <30 mL/min) or patient on dialysis
21. Planned treatment with another investigational device or procedure during the study period
22. Balloon valvuloplasty (BAV) within 30 days of the procedure
23. Any planned surgical or interventional cardiac procedure (e.g., concurrent coronary revascularization or AF ablation) during the TAVR procedure, within 30 days before or after the TAVR procedure
24. Emergency surgery for any reason
25. Pregnancy, lactation or intent to become pregnant during study participation
26. Unable or unwilling to complete all required screening and/or follow-up assessments, including subjects with active major psychiatric disease; with severe visual, auditory, or learning impairment
27. Investigator considers participation in the study not to be in the subject's best interest
28. Dementia or any other cognitive deficit that results in inability to provide informed consent or comply with the study protocol
29. Presence of hemodialysis shunt, graft, or arterio-venous fistula involving access vasculature

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority | Non-inferiority of 30-day Emboliner device MACCE patient incidence rate compared to the Sentinel device patient incidence rate.
  Non-inferiority of 30-day Emboliner device MACCE patient incidence rate compared to the Sentinel device patient incidence rate.
  K4: Description Non-inferiority of 30-day Emboliner device MACCE patient incidence rate compared to the Sentinel device patient incidence rate.
  30 Days

SECONDARY OUTCOMES:
Non-inferiority VARC-2 | 30 Days
  Non-inferiority of 30-day Emboliner device VARC 2-defined stroke incidence rate compared to the Sentinel device incidence rate.
Debris Capture | 30 Days
  The count (by number of particles >150 microns) of debris capture using the Emboliner device will be compared to the count of debris captured by the Sentinel device.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Brenton, Study Director — Emboline, Inc.
Locations (2):
- United States (2):
  - NewYork-Presbyterian/Columbia University Medical Center, New York, New York
  - Oklahoma Heart Institute, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No